CLINICAL TRIAL: NCT05011760
Title: [C-11]NPA PET-amphetamine in Cocaine Use Disorders (Aim 2)
Brief Title: [C-11]NPA PET-amphetamine in Cocaine Use Disorders
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Rajesh Narendran (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor-Investigator, Rajesh Narendran, Professor of Radiology and Psychiatry, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: STUDY20060171 (Aim 2); R01DA026472 (NIH)
Record Dates: First submitted 2021-08-11; First posted 2021-08-18 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-06

CONDITIONS: Cocaine Use Disorder
Keywords: [C-11]NOP-1A, [C-11]NPA , nociceptive opioid peptide receptors, dopamine release
MeSH Terms: interventions — BaseLine dental cement; Dextroamphetamine

STUDY DESIGN:
Intervention Model Description: Single group, correlational analyses
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- PET (Experimental): [C-11]NPA PET Scan
  Interventions: Radiation: Baseline [C-11]NPA PET Scan; Drug: d-amphetamine; Radiation: Post-amphetamine [C-11]NPA PET Scan

INTERVENTIONS:
Radiation: Baseline [C-11]NPA PET Scan — Radiotracer
Drug: d-amphetamine — Oral, 0.5 mg/Kg
Radiation: Post-amphetamine [C-11]NPA PET Scan — Radiotracer

SUMMARY:
This study uses [11C]NPA positron emission tomography (PET) and a d-amphetamine challenge to image amphetamine induced dopamine release in the striatum in subjects with cocaine use disorders (CUD). Amphetamine-induced dopamine release data from this study will be correlated with [11C]NOP-1A VT measured at baseline in the midbrain. [11C]NOP-1A PET data will be used from aim 1 (see, Study Record: Imaging CRF X NOP interactions in Cocaine Use Disorders)

DETAILED DESCRIPTION:
Cocaine use disorder (CUD) is a chronic disorder associated with numerous relapses and periods of abstinence.

Studies in CUD suggest that ~ 60 to 75% of abstinent addicts relapse over twelve months. Documenting specific neurochemical abnormalities that lead to relapse in individuals with CUD has the potential to accelerate the development of medications to prevent relapse. Basic investigations postulate an imbalance between brain stress and anti-stress/resilience systems as the underlying mechanism that drives negative reinforcement, craving, and relapse in addiction.. Nociceptin (N/OFQ), which binds to the nociceptive opioid peptide receptors (NOP) is a critical component of the brain's anti-stress system. N/OFQ exerts its anti-stress effect by counteracting the functional effects of the primary stress-promoting neuropeptide corticotrophin releasing factor (CRF) in the brain. Studies have also shown that acute increases in CRF and stress are countered by increased NOP receptor expression (~ 10% ) in brain regions that regulate stress such as bed nucleus of the stria terminalis. PET studies with the NOP radiotracer [11C]NOP-1A show increased binding to NOP in CUD compared to HC. PET studies also show NOP receptors to upregulate (~ 15%) in response to an acute intravenous hydrocortisone challenge (1 mg/Kg). NOP upregulation may represent an adaptive mechanism in the brain to counteract stress-induced increases in cortisol and CRF. Here, we postulate a failure in this adaptive mechanism as a reason that leads to relapse in CUD. CUD subjects and HC will be studied with [11C]NOP-1A before and after an intravenous hydrocortisone challenge (aim 1). Hydrocortisone is used as a challenge because it increases cortisol and CRF in brain regions that regulate stress. We hypothesize that hydrocortisone-induced increases in [11C]NOP-1A binding (DELTA VT) will be smaller in CUD relative to HC, and this will be associated with less time to relapse in a 12-week follow up. Mechanistic studies have also shown N/OFQ to act on ventral tegmental area/midbrain NOP receptors to inhibit the firing of dopamine neurons and limit reward to cocaine. Imaging amphetamine-induced dopamine release in a subset of CUD subjects who participate in aim 1 will allow us to link midbrain NOP receptor expression with ventral striatum (VST) dopamine release and examine its role in reinforcement (aim 2). The aims proposed in this study have the potential to clarify the role of N/OFQ and NOP in stress, reward, and relapse in CUD.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females between 18 and 55 years old
2. Fulfil DSM-5 criteria for cocaine use disorder
3. No other current DSM-5 psychiatric or addictive disorders (such as major depressive disorder, bipolar disorders, psychotic disorders, etc.,)
4. No current abuse (six months) of opiates, sedative-hypnotics, amphetamines, and MDMA as well as moderate to severe alcohol or cannabis use (twice a week). Nicotine use will be quantified and controlled between groups using the Fagerstrom Test for Nicotine Dependence (Heatherton et al., 1991);
5. Not currently on prescription medical or psychotropic medications
6. No current or past severe medical, endocrine or neurological illnesses including glaucoma, seizure disorders, hypertension, hypercholesterolemia as assessed by a complete medical history and physical
7. Not currently pregnant or breastfeeding
8. No history of significant radioactivity exposure in past year from another research study or occupation that exceeds RDRC guidelines
9. No metallic objects in the body that are contraindicated for MRI
10. No baseline BP ≥ 140/90 and/or HR ≥ 100.
11. No first-degree relative with an MI or stroke prior to middle age
12. No first-degree relative with psychosis or mania.
13. Completed a baseline [11C]NOP-1A PET scan in Aim 1 (Study Record: Imaging CRF X NOP interactions in Cocaine Use Disorders)

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-01-31 (Actual); Primary Completion 2028-09-01 (Estimated); Study Completion 2028-09-01 (Estimated)

PRIMARY OUTCOMES:
DELTA binding potential relative to non displaceable uptake (BPND) | Baseline, and 2.5 to 3 hours post-amphetamine
  DELTA BPND is the change in BPND from the baseline PET scan to post-amphetamine PET scan that will be acquired 2.5 to 3 hours after d-amphetamine administration (0.5 mg/Kg, oral)

CONTACTS AND LOCATIONS:
Overall Officials: Rajesh Narendran, Principal Investigator — University of Pittsburgh
Locations (1):
- University of PIttsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No